CLINICAL TRIAL: NCT00428181
Title: Multidisciplinary Approach to Reduce Injury and Alcohol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Craig Field, Ph.D., Principal Investigator, University of Texas at Austin
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA_FIE_015439; R01AA015439 (NIH); NIH Grant 1R01 AA015439
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Drinking Behavior; Injury Recidivism
Keywords: Brief alcohol intervention; Booster session; Personalized feedback; Motivational interview; Injury recidivism; Psychological Interview; Risk Reduction Behaviors
MeSH Terms: conditions — Drinking Behavior; Risk Reduction Behavior | interventions — Ethanol; Methods; Immunization, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Brief Intervention (Active Comparator): The primary purpose of the proposed research is to compare the effectiveness of brief intervention, brief intervention plus a booster and treatment as usual for adult patients with an alcohol related injury.
  Interventions: Behavioral: Brief alcohol intervention
- 2) Booster (Active Comparator): The primary purpose of the proposed research is to compare the effectiveness of brief intervention, brief intervention plus a booster and treatment as usual for adult patients with an alcohol related injury.
  Interventions: Behavioral: Brief alcohol intervention plus booster

INTERVENTIONS:
Behavioral: Brief alcohol intervention — Brief alcohol intervention
  Arms: 1 Brief Intervention
Behavioral: Brief alcohol intervention plus booster — Brief alcohol intervention plus booster in a later session
  Arms: 2) Booster

SUMMARY:
The purpose of this study is to determine whether a booster session is needed after a brief intervention upon initial admission to the emergency room (ER) in order to reduce the rate of alcohol-related injury recidivism.

DETAILED DESCRIPTION:
The primary purpose of the proposed research is to compare the effectiveness of brief intervention, brief intervention plus a booster and treatment as usual for adult patients with an alcohol related injury. The primary outcomes of interest in the proposed trial are injury recidivism, alcohol intake, and alcohol problems. Because brief alcohol interventions with injured patients are opportunistic in nature, the patient's motivation to change or stage of change likely influences their response to brief intervention as well as the need for additional intervention. Therefore, the primary hypothesis of the proposed research is that patients presenting for treatment of an alcohol related injury who are in the precontemplation or contemplation stages of change require brief intervention with booster while patients in the preparation or action stages of change benefit equally from brief intervention alone or brief intervention plus booster. That is, an interaction between the patient's stage of change (Precontemplation and Contemplation or Action) at enrollment and treatment type (Brief Intervention, Brief Intervention with Booster and Treatment as Usual) is hypothesized to influence treatment effect at follow up. In addition, the impact of intervention on the patient's motivation to change at follow up will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated for an intentional or unintentional injury associated with motor vehicle collisions involving driver (i.e., passenger or pedestrian) will be eligible for inclusion in the study.
* Patients who are treated for an intentional or unintentional injury associated with violence-related injuries including gunshot wounds, stab wounds, or other injuries related to assaults and falls will be eligible for inclusion in the study.
* Patients must be eighteen years of age or older.
* Study clinicians actively monitor these patients on a daily basis and the patient's ability to participate is determined through the use of hospital medical records, daily contact with the emergency department nursing staff and hospital personnel as well as direct contact with the patient.
* Currently, patients who are intoxicated at the time of admission to the emergency room are maintained in an observation area or admitted for twenty-three hour observation in order to rule out severe injury. They will be monitored by study personnel on an hourly basis and approached to participate in the study after evidence of acute intoxication has subsided.
* Admitted patients who are intoxicated will be approached during their hospital stay after they are medically stable.

Exclusion Criteria:

* Patients with other penetrating trauma not related to motor vehicle collisions, violence or falls, such as poisoning, bites, contusions, concussions, strains and sprains are excluded.
* Patients with traumatic brain injury, or a Glasgow Coma Scale (GCS) score of less than 15, are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Reduction in injury recidivism | August 2011
Reduction in alcohol intake | August 2011
Reduction in alcohol problems | August 2011

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Field, PhD, Principal Investigator — UT Austin School of Social Work
Locations (3):
- United States (3):
  - Brackenridge University Medical Center, Austin, Texas
  - Methodist Health System, Dallas, Texas
  - Baylor University Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Derived] Cochran G, Field C, Foreman M, Ylioja T, Brown CV. Effects of brief intervention on subgroups of injured patients who drink at risk levels. Inj Prev. 2016 Jun;22(3):221-5. doi: 10.1136/injuryprev-2015-041596. Epub 2015 Jun 29. PMID 26124071
- [Derived] Field C, Walters S, Marti CN, Jun J, Foreman M, Brown C. A multisite randomized controlled trial of brief intervention to reduce drinking in the trauma care setting: how brief is brief? Ann Surg. 2014 May;259(5):873-80. doi: 10.1097/SLA.0000000000000339. PMID 24263324